CLINICAL TRIAL: NCT05337267
Title: Phase I Study to Evaluate PK Similarity of Recombinant Fully Human Anti-programmed Death Receptor 1 Monoclonal Antibody Injection Before and After IBI308 Manufacturing Process Change in Healthy Chinese Male Subjects
Brief Title: Phase I Study of Sintilimab in Healthy Chinese Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: CIBI308K102
Record Dates: First submitted 2022-03-22; First posted 2022-04-20 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2022-12

CONDITIONS: Healthy Male Subjects
MeSH Terms: interventions — sintilimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sintilimab (after the change) (Experimental)
  Interventions: Drug: sintilimab (before the change)
- sintilimab (before the change) (Active Comparator)
  Interventions: Drug: sintilimab (after the change)

INTERVENTIONS:
Drug: sintilimab (after the change) — 0.3mg/kg，I.V.，single dose
  Arms: sintilimab (before the change)
Drug: sintilimab (before the change) — 0.3mg/kg，I.V.，single dose
  Arms: sintilimab (after the change)

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetic similarity of sintilimab with different manufacturing process in healthy male subjects. Another purpose is to determine safety, and immunogenicity of sintilimab with different manufacturing process，also to determine Pharmacodynamics of sintilimab with different manufacturing process in 12 healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Males aged 18 to 45 (including both ends);
2. Body Mass Index (BMI) is 19.0~28.0 kg/m2 (including both ends), and body weight is 62.0~73.0kg (including both ends);
3. The investigator is assessed as a healthy male subject based on a complete medical history, including physical examination, vital signs, 12-lead electrocardiogram and laboratory tests;
4. Subjects agree to use reliable contraceptive measures (such as abstinence, sterilization, contraceptives, injectable contraceptive medroxyprogesterone or subcutaneous implant contraception, etc.) during the study period and within 6 months after the study drug infusion. );
5. Fully understand the purpose of the trial, understand the pharmacological effects of the study drug and possible adverse reactions; and abide by the trial process and voluntarily sign the informed consent.

Exclusion Criteria:

1. Those with a history of chronic liver, kidney, cardiovascular, neurological/mental, digestive tract, respiratory, urinary, endocrine and other systemic diseases;
2. Those with a history of autoimmune diseases (see Annex 1);
3. Regular drinkers within 6 months prior to screening (regular drinkers are defined as drinking more than 2 units per day on average, or drinking more than 14 units per week on average: 1 unit = 360ml of beer or 45ml of alcohol for 40 % above spirits or 150ml wine);
4. Subjects who have had opportunistic infections within 6 months before screening (such as: herpes zoster, active cytomegalovirus, Pneumocystis carinii, histoplasma, aspergillus, mycobacteria, etc. );
5. Known history of recurrent or chronic infection, history of chronic or recurrent infection, including but not limited to: chronic kidney infection, chronic chest infection (such as bronchiectasis), sinusitis, recurrent urinary tract infection, Open, draining or infected skin wounds;
6. Those with a history of acute infection within 2 weeks before screening;
7. A history of malignant tumor, unless it is a skin squamous cell carcinoma or basal cell carcinoma that has been successfully resected and has no evidence of metastasis;
8. Those who are suspected or confirmed to be allergic or have had severe drug or food allergy reactions in the past, have a clear history of allergies and/or are allergic to the study drug or its components after inquiries;
9. Have used any drugs (including traditional Chinese medicines and vitamins) within 2 weeks before screening, or the last medication is less than 5 half-lives of the drug from the test administration day, whichever is longer;
10. Those who have used anti-PD-1/PD-L1 drugs in the past;
11. Those who have participated in other interventional clinical trials within 3 months before screening;
12. Those who lost blood, donated blood or received any blood product transfusion of ≥400 ml within 3 months before screening;
13. Those who received major surgery or hospitalization due to illness within 3 months before screening;
14. Those who have been vaccinated with live vaccines within 6 months before screening, or who are expected to receive live vaccines during the study period;
15. Those with a history of drug abuse or positive drug screening results within 12 months before screening;
16. Those with abnormal vital signs and physical examination during the screening period and judged by the research doctor to have clinical significance;
17. Abnormal electrocardiogram (such as QTcF>450ms, shortened or prolonged PR interval, second-degree and third-degree atrioventricular block, pre-excitation syndrome, etc.) during the screening period and judged by the research doctor to be clinically significant;
18. Abnormal chest X-ray (frontal and lateral) or lung CT during the screening period and judged by the research doctor to have clinical significance;
19. Abnormal laboratory tests and clinical significance during the screening period. (Remarks: If there is any abnormality and it has clinical significance as judged by the research doctor, if it is within the normal range after re-examination, it can also be included in the group);
20. Patients with known history of tuberculosis or suspected clinical manifestations of tuberculosis (including but not limited to pulmonary tuberculosis, lymph node tuberculosis, tuberculous pleurisy, etc.), positive test for tuberculosis laboratory test (QuantiFERON-TB tuberculosis test/T.SPOT tuberculosis test) examinee;
21. Human Immunodeficiency Virus (HIV) antibody, Hepatitis C virus (HCV) antibody, syphilis test (RPR), Hepatitis B virus (HBV) surface antigen, e antigen ( Positive results for either HBeAg) or core antibody (HBcAb);
22. Subjects who have a reproductive plan from the screening period to 6 months after the administration of the study drug, or who are unwilling to take the contraceptive measures specified in the protocol during the trial;
23. The investigator believes that it is not suitable to participate in this clinical trial due to other reasons.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Age≥18 years and ≤45 years, healthy male subjects
Enrollment: 117 (Actual)
Dates: Start 2022-04-13 (Actual); Primary Completion 2023-05-24 (Actual); Study Completion 2023-07-24 (Actual)

PRIMARY OUTCOMES:
Pre-experiment: Treatment-emergent Adverse Events (TEAEs) graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0 (NCI-CTCAE v5.0) incidence. | Day 43
Pre-experiment: Serious Adverse Events (SAEs) graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0 (NCI-CTCAE v5.0) incidence. | Day 43
Formal test: Bioequivalence results using the area under the plasma concentration-time curve (AUC0-inf) as the judging indicators. | Day 57
Bioequivalence results using the peak serum drug concentration (Cmax) as the judging indicators. | Day 57

SECONDARY OUTCOMES:
Other PK parameters: Area under the plasma concentration-time curve (AUClast) | Day 57
Other PK parameters: Volume of distribution (V) | Day 57
Other PK parameters: Clearance (CL) . | Day 57
Other PK parameters: Half-life (t1/2). Other PK parameters, including but not limited to elimination half-life (t1/2). | Day 57
The occurrence of Neutralizing antibodies Antibody(NAb) | Day 57
The occurrence of Anti-drug Antibody(ADA) | Day 57
PD indicator: PD-1 receptor occupancy rate. | Day 57

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Cancer Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No